CLINICAL TRIAL: NCT01456403
Title: Histological Validation Of Carotid Plaque Composition In Preoperative Imaging Of Patients Scheduled For Carotid Endarterectomy
Brief Title: Histological Validation Of Carotid Plaque Composition In Preoperative Imaging
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, J. David Spence, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: CAIN-002
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Carotid Stenosis
Keywords: Carotid; endarterectomy; vulnerable plaque; Ultrasound; MRI; PET/CT
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Histological sections
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Carotid endarterectomy patients: Patients scheduled for clinically indicated carotid endarterectomy
  Interventions: Other: Histological validation

INTERVENTIONS:
Other: Histological validation — 3D ultrasound, PET/CT, MRI, contrast ultrasound

SUMMARY:
Patients scheduled for carotid endarterectomy undergo preoperative imaging to assess vulnerable plaque. The imaging modalities include (in various combinations at different study sites) 3-dimensional ultrasound, PET/CT imaging with fluorodeoxyglucose, MRI (3T)with gadolinium, and contrast ultrasound for assessment of neovascularity of plaques. At surgery the carotid endarterectomy is carried out with en bloc removal of the specimen, which is scanned and stained and assembled into 3D histology.

DETAILED DESCRIPTION:
Detailed Description: Patients will undergo 3D U/S and at least one other imaging method, PET/CTA or MRI, preoperatively. At some sites, some patients will also have an ultrasound with microbubbles. Following surgery, the carotid specimens will be transported to a central pathology lab for microcomputed tomographic imaging and further study.

At some sites patients will have a follow-up 3D U/S approximately 1 year after surgery to determine progression of plaque.

CAIN-2 sub-studies:

Eligible patients may be enrolled into one of the following sub-studies:

1. CAIN-2 NaF pilot Characterizing Atherosclerotic Plaque with Sodium Fluoride Positron Emission Tomography- A Sub-Study of the Canadian Atherosclerosis Imaging Network (CAIN Project 2), - patients undergo sodium fluoride (NaF) PET/CT with CTA instead of FDG PET/CT preoperatively. All other imaging and study procedures are carried out as per the CAIN-2 study.

   Recruitment for this pilot study is complete.
2. CAIN-2B Atherosclerotic plaque imaging using NaF and FDG imaging: Validation and Evaluation of Disease Progression. A sub-study of the Canadian Atherosclerosis Imaging Network (CAIN-2) Histopathology Validation study - patients undergo both NaF and FDG PET/CT preoperatively. All other imaging and study procedures are carried out as per the CAIN-2 study.

A total of 45 patients will be enrolled in this sub-study. Eligibility criteria for the sub-studies is identical to the CAIN-2 criteria.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for carotid endarterectomy; provided informed consent

Exclusion Criteria:

* Those not eligible for some of the imaging modalities (for example, metal in body, renal dysfunction) are excluded from MRI imaging or CT angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for carotid endarterectomy
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2011-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Histologic validation of preoperative imaging of vulnerable plaque | Cross-sectional
  3D histological images registered to the preoperative images of carotid plaques will be used to validate imaging features of plaque such as thin cap, intraplaque hemorrhage, large lipid core and inflammation.

SECONDARY OUTCOMES:
Prediction of cardiovascular events | 2 years
  Occurrence of stroke, cardiovascular death, myocardial infarction or revascularization procedures by imaging features of vulnerable plaque in the baseline images

CONTACTS AND LOCATIONS:
Overall Officials: J. David Spence, M.D., Study Chair — Robarts Research Institute, University of Western Ontario
Locations (3):
- Canada (3):
  - Robarts Research Institute, London, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Does Glucose Corrected [18F]fluorodeoxyglucose Uptake in Human Carotid Plaque Relate to the Extent of Inflammation on Immunohistology? Cocker M.S., Spence J.D., Hammond R., Mc Ardle B., deKemp R., Brennan J., Lum C., Yerofeyeva Y., Karavardanyan T., Adeeko A., Youssef G., Hill A., Stotts G., Renaud J.M., Alturkustani M., Hammond L., DaSilva J., Tardif J.C. and Beanlands R. American Heart Association Scientific Sessions. Los Angeles, United States. November 3 - 7, 2012. Circulation 2012: 126: A17612.
- [Background] Immunohistochemical Validation of [18F]-fluorodeoxyglucose as a Novel Biomarker of Inflamed Vulnerable Carotid Plaque: A Sub-study of the Canadian Atherosclerosis Imaging Network (CAIN). Cocker M.S., Mc Ardle B., deKemp R., Lum C., Youssef G., Hammond R., Yerofeyeva Y., Karavardanyan T., Adeeko A., Hill A., Stotts G., Sharma M., Renaud J.M., Brennan J., Alturkustani M., Hammond L., DaSilva J., Tardif J.C. Spence J.D., and Beanlands R. Canadian Cardiovascular Congress 2012. Toronto, Canada. October 26 - 31, 2012. Canadian Journal of Cardiology 2012: 28(5): S162.
- [Result] Cocker MS, Mc Ardle B, Spence JD, Lum C, Hammond RR, Ongaro DC, McDonald MA, Dekemp RA, Tardif JC, Beanlands RS. Imaging atherosclerosis with hybrid [18F]fluorodeoxyglucose positron emission tomography/computed tomography imaging: what Leonardo da Vinci could not see. J Nucl Cardiol. 2012 Dec;19(6):1211-25. doi: 10.1007/s12350-012-9631-9. PMID 23073913
- See also: CAIN website — http://www.canadianimagingnetwork.org/